CLINICAL TRIAL: NCT00971893
Title: A Prospective Study to Assess the Safety and Effectiveness of Medrol® in Acute Asthma in Indian Patients
Brief Title: A Study To Assess The Safety And Effectiveness Of Medrol® In Acute Asthma In Indian Patients
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0121003
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Asthma
Keywords: Acute Exacerbation of Bronchial Asthma Acute Asthma
MeSH Terms: conditions — Asthma | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methylprednisolone Group
  Interventions: Drug: Oral Methylprednisolone Tablets

INTERVENTIONS:
Drug: Oral Methylprednisolone Tablets — Oral Methylprednisolone tablets given as per locally approved prescribing information

SUMMARY:
The present study is designed to collect data on real world experience on use of Medrol in acute asthma in Indian patients.

DETAILED DESCRIPTION:
Sequential enrollment

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrollment in this study, patients must be prescribed oral Medrol® tablets (4mg and 16 mg) for acute asthma as per the locally approved prescribing information. The prescription of Medrol® will be separated from the decision to include the patient in the study.
* Medrol® tablets, will be prescribed to the patient by the physician according to his/her usual practice. The decision to prescribe Medrol® tablet will necessarily precede and will be independent of the decision to enroll patient into the study. Only those patients who have been prescribed Medrol® tablets will be evaluated for their potential eligibility for the study
* Only those patients, who are ready and willing to sign an informed consent, will be included in the study
* Subject can be contacted through telephone

Exclusion Criteria:

* Based upon history or physical exam in the emergency department (ED) or Clinic, subjects with known or suspected cause of pulmonary symptoms other than asthma, such as COPD, CHF, pneumonia, pulmonary embolism, or angioedema
* Any contraindication to Medrol tablet use. Contraindications of Medrol use are systemic fungal infections and known hypersensitivity to components

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of Acute Asthma who have been prescribed oral Medrol tablets, will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Relapse within 10 days of hospital discharge (Relapse is defined as unscheduled care at a doctor's office, a clinic, or Emergency Department (ED) for symptoms of persistent or worsening asthma after hospital discharge) | 10 days after discharge

SECONDARY OUTCOMES:
Relapse within 20 days of hospital discharge (Relapse is defined as above for Primary Endpoint). | 20 days after discharge
Change in PEFR (Peak Expiratory Flow Rate measured in Percentage of expected) between start of therapy and first follow up visit. | 8 - 22 days after discharge
Change in FEV1 (Forced Expiratory Volume in 1 second) between start of therapy and first follow up visit. | 8 - 22 days after discharge
Proportion of patients controlled for asthma symptoms in the last 7 days after 10 days of hospital discharge | 10 days after discharge
Proportion of patients controlled for asthma symptoms in the last 7 days after 20 days of hospital discharge | 20 days after discharge
Change in frequency in last 24 hours of inhalational Beta 2 agonist therapy between start of therapy and first follow up visit | 8 - 22 days after discharge
Physician-directed intensification of pharmacologic therapy between discharge from hospital and first follow up visit. | 8 - 22 days after discharge
Summary of adverse events in the study | Baseline to 20 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0121003&StudyName=A%20Study%20To%20Assess%20The%20Safety%20And%20Effectiveness%20Of%20Medrol%AE%20In%20Acute%20Asthma%20In%20Indian%20Patients